CLINICAL TRIAL: NCT00874003
Title: The Effects of Mirtazapine vs Placebo on Alcohol Consumption in Male Alcohol High Consumers; a Randomized Controlled Trial
Brief Title: The Effects of Mirtazapine Versus Placebo on Alcohol Consumption in Male Alcohol High Consumers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Bo Söderpalm/ MD, PhD, sponsor, Addiction Biology Unit, Sahlgrenska University Hospital, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOTABU-BO1
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-03

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; anti-depressant; 5-HT; NE
MeSH Terms: conditions — Alcoholism | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mirtazapine, tablet, 30 mg (Experimental): n=29
  Interventions: Drug: mirtazapine
- sugar pill (Placebo Comparator): n=30
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mirtazapine — oral tablet, 30 mg daily
  Arms: mirtazapine, tablet, 30 mg
Drug: placebo — oral tablet, 1 daily
  Arms: sugar pill

SUMMARY:
The purpose of this study is to study the effects of 8 weeks of treatment with mirtazapine on alcohol consumption in alcohol high consuming men. This study is a randomized, double-blind placebo controlled clinical trial with parallel group design(N=59).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* male sex
* alcohol high consumption
* signed informed consent

Exclusion Criteria:

* psychiatric disorders (except nicotine and alcohol dependence)
* severe somatic disorders
* inadequate knowledge of the Swedish language

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-04; Primary Completion 2006-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption measured by alcohol diary (units/week).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea deBejczy, MD, Study Director — Addiction Biology Unit; Bo Söderpalm, MD, PhD, Principal Investigator — Addiction Biology Unit
Locations (1):
- Addiction Biology Unit, Gothenburg, Sweden